CLINICAL TRIAL: NCT07196566
Title: Double-Layer Closure of Oroantral Fistula Using Buccal Split-Thickness and Palatal Subepithelial Connective Tissue Flaps
Brief Title: Double-Layer Closure Technique Using Buccal and Palatal Flaps for Oroantral Fistula
Acronym: OAF-DLC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed sobhie abdelhameed, Teaching assistant in oral and maxillofacial department, faculty pf dentistry, Tanta university, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TantaOMS-OAF-DLC2025
Record Dates: First submitted 2025-09-12; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Oroantral Fistula; Double Layer
Keywords: oroantral fistula; double layer closure; buccal flap; palatal flap; rotational palatal connective tissue flap
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Intervention Model Description: All enrolled patients will undergo closure of chronic oroantral fistula using double-layer technique consist of split thickness buccal, palatal flap and rotational palatal underlaying connective tissue.
  this a single-arm, prospective clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Double-Layer Closure of Oroantral Fistula Using Buccal and palatal Split-Thickness flap (Experimental): A prospective clinical case series was conducted involving twelve patients with oroantral fistulas ≥5 mm in diameter. Closure was performed using split-thickness buccal and palatal mucosal flaps with a subepithelial palatal connective tissue graft rotated to cove the bony defect and sutured to the buccal periosteum as the first layer, then the buccal mucosa sutured with the palatal one . Clinical evaluations were conducted at regular intervals over a 3-month postoperative period, assessing wound healing, fistula recurrence, pain, facial edema, infection, and donor site morbidity.
  Interventions: Procedure: Closure was performed using split-thickness buccal and palatal mucosal flaps with a subepithelial palatal connective tissue graft

INTERVENTIONS:
Procedure: Closure was performed using split-thickness buccal and palatal mucosal flaps with a subepithelial palatal connective tissue graft — Closure was performed using split-thickness buccal and palatal mucosal flaps with a subepithelial palatal connective tissue graft rotated to cove the bony defect and sutured to the buccal periosteum as the first layer, then the buccal mucosa sutured with the palatal one . Clinical evaluations were conducted at regular intervals over a 3-month postoperative period, assessing wound healing, fistula recurrence, pain, facial edema, infection, and donor site morbidity.

SUMMARY:
A prospective clinical case series was conducted involving twelve patients with oroantral fistulas ≥5 mm in diameter. Closure was performed using split-thickness buccal and palatal mucosal flaps with a subepithelial palatal connective tissue graft rotated to cove the bony defect and sutured to the buccal periosteum as the first layer, then the buccal mucosa sutured with the palatal one . Clinical evaluations were conducted at regular intervals over a 3-month postoperative period, assessing wound healing, fistula recurrence, pain, facial edema, infection, and donor site morbidity.

DETAILED DESCRIPTION:
The proposed double-layer technique achieved high success rates in closing oroantral fistulas with minimal postoperative complications, reduced facial edema, and better preservation of vestibular depth compared to conventional techniques.

A prospective clinical case series was conducted involving twelve patients with oroantral fistulas ≥5 mm in diameter. Closure was performed using split-thickness buccal and palatal mucosal flaps with a subepithelial palatal connective tissue graft rotated to cove the bony defect and sutured to the buccal periosteum as the first layer, then the buccal mucosa sutured with the palatal one . Clinical evaluations were conducted at regular intervals over a 3-month postoperative period, assessing wound healing, fistula recurrence, pain, facial edema, infection, and donor site morbidity.

This technique demonstrated reliable, tension-free closure with excellent clinical outcomes, reduced postoperative facial edema, and preserved vestibular depth, supporting its potential as an effective and safe surgical option for managing oroantral fistulas.

The purpose of the present study was explained to the patients and informed consents were obtained according to the guidelines on human research adopted by the Research Ethics Committee, Faculty of Dentistry, Tanta University.

ELIGIBILITY:
Inclusion Criteria:

* patients with oroantral fistula

Exclusion Criteria:

* patients with repeated oroantral fistula closure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
recurrence of fistula | one week -4 weeks
  presence of oroantral fistula or not
vestibular height | 1-3 months postoperatively
  using periodontal prob

CONTACTS AND LOCATIONS:
Overall Officials: mohamed s abdelhameed, Asst lecturer, Principal Investigator — Tanta University
Locations (1):
- faculty of dentistry, Tanta university, Tanta, Egypt